CLINICAL TRIAL: NCT02237885
Title: Pain Management Using Mobile Technology in Veterans With PTSD and TBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: Pro00068864; R34AT008399-01 (NIH); 14-1138 (Other: University of North Carolina - Chapel Hill); Pro00068864 (Other: Duke University Health System IRB)
Record Dates: First submitted 2014-09-09; First posted 2014-09-11 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Chronic Pain; Posttraumatic Stress Disorders; Traumatic Brain Injury
Keywords: Military Veterans
MeSH Terms: conditions — Chronic Pain; Stress Disorders, Post-Traumatic; Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Neurofeedback (Experimental)
  Interventions: Device: NeuroSky MindWave Mobile

INTERVENTIONS:
Device: NeuroSky MindWave Mobile
  Other Names: Mobile Neurofeedback (Application); Apple iPod touch

SUMMARY:
Up to half of military veterans with traumatic brain injury (TBI) also suffer from co-occurring posttraumatic stress disorder (PTSD). Both are linked to higher risk of chronic pain, one of the most common health complaints among U.S. veterans who served in Operation Enduring Freedom (Afghanistan), Operation Iraqi Freedom (Iraq), and Operation New Dawn (OEF/OIF/OND). However, pain medications elevate risk of opioid abuse, and studies indicate that veterans perceive barriers to traditional mental health treatments. Little research exists regarding non-pharmacological, technology-based interventions designed to reduce pain in veterans with PTSD and TBI. Mobile technology used to implement neurofeedback (EEG biofeedback) shows promise in providing a portable, low-cost intervention for reducing pain in veterans with co-occurring disorders. We aim to test the feasibility and effectiveness of using mobile neurofeedback devices for reducing pain symptoms in veterans with PTSD and TBI. Veterans with PTSD, TBI, and chronic pain will receive a NeuroSky headset (which reads EEG brain waves) and an iPod Touch with an app called Mobile Neurofeedback (which provides neurofeedback to induce relaxation). Veterans are taught how to use these together to do neurofeedback themselves at home for 12 weeks. Guided by existing research and preliminary data, we hypothesize that participants will show high levels of adherence to the NeuroSky + Mobile Neurofeedback intervention for the 3-month study duration and that participants will show statistically significant reduction in pain symptoms at 3 months compared to baseline. Given links between pain and other outcomes in veterans, we will also explore effects on drug abuse, violence, and suicidality. When the research is complete, the field will be changed because we will know whether new technology reading EEG brainwaves can be used to treat symptoms among individuals suffering from chronic pain. We will also know whether neurofeedback shows promise as an effective intervention for veterans with PTSD and TBI to reduce pain and related outcomes. If this program of research is successful, its impact will be to shift approaches to managing pain in clinical practice, for both veterans and civilians

ELIGIBILITY:
Inclusion Criteria:

* Military veteran who served during Operation Enduring Freedom (OEF), Operation Iraqi Freedom (OIF), and/or Operation New Dawn (OND)
* Posttraumatic Stress Disorder (PTSD)
* Traumatic Brain Injury (TBI)
* Chronic pain

Exclusion Criteria:

* History of epilepsy, seizure disorder, or have ever had a seizure or epileptic fit
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2017-11-21 (Actual); Study Completion 2017-11-21 (Actual)

PRIMARY OUTCOMES:
Number of ten minute neurofeedback sessions completed on mobile platform | 3 months
  Per protocol, participants will be requested to complete 4 neurofeedback sessions per week for 12 weeks. This data will be collected on participants' mobile devices.

SECONDARY OUTCOMES:
Change in participant's self-reported pain score from 0-10, 0 least amount of pain, 10 highest | Baseline, 3 months
  Per protocol, participants are enrolled if they have chronic pain defined as self-reporting on the numeric rating scale a score of 4 or above lasting three months or more. The study will therefore ask participants to self report their level of pain (from 0-10, 0 least amount of pain, 10 being the most) following the three months of the neurofeedback sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Elbogen, PhD, Principal Investigator — Duke University, Dept. of Psychiatry
Locations (1):
- Duke University, Department of Psychiatry, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Elbogen EB, Alsobrooks A, Battles S, Molloy K, Dennis PA, Beckham JC, McLean SA, Keith JR, Russoniello C. Mobile Neurofeedback for Pain Management in Veterans with TBI and PTSD. Pain Med. 2021 Feb 23;22(2):329-337. doi: 10.1093/pm/pnz269. PMID 31697371